CLINICAL TRIAL: NCT02572895
Title: Recurrent Urinary Tract Infection Prevention With Biologic Cranberry Extract Intake Standardized in Proanthocyanidins: A Double-blind Clinical Trial
Brief Title: Cranberry Extract and Urinary Infection Prevention: a Clinical Trial
Acronym: PACCANN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Ministry of Agriculture, Fisheries and Food, Quebec (Other Government); Nutra Canada (Other)
Responsible Party: Principal Investigator, Sylvie Dodin, MD, M.Sc., Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PACCANN_2015
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Tract Infections
Keywords: Cranberry; Proanthocyanidins; Urinary catabolites
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimal dose (Active Comparator): One capsule with a proanthocyanidins standardized cranberry extract of 18,5 mg twice a day, i.e. in the morning and at night.
  Interventions: Dietary Supplement: Cranberry extract
- Control dose (Placebo Comparator): One capsule with a proanthocyanidins standardized cranberry extract of 1 mg twice a day, i.e. in the morning and at night.
  Interventions: Dietary Supplement: Cranberry extract

INTERVENTIONS:
Dietary Supplement: Cranberry extract — The aim of this clinical trial is to assess efficacy of an optimal dose of cranberry extract compared to a control dose on mean number of new UTIs for a 6-month period follow-up in women. Participants will be randomly assigned to the optimal dose or control dose treatment at their first visit at the Institute of Nutrition and Functional Foods. This intervention includes three visits at 0, 12 and 24 weeks. At the first visit, women will have to complete questionnaires to provide sociodemographic, medication and natural health products, health antecedents and quality of life information and to document risk factors related to UTIs. A 24-hour recall questionnaire about consumption of PACs will also be completed. A urinary sample analysis and culture as well as a pregnant test will also be performed. Compliance regarding capsules' intake and potential side effects will be documented. The completion of questionnaires and urinary measurements will be repeated at weeks 12 and 24.

SUMMARY:
The purpose of this clinical trial study is to assess, among young and sexually active women presenting recurrent urinary tract infection (UTIs), efficacy of an optimal dose of cranberry extract quantified and standardized to 37 mg/day of Proanthocyanidins (PACs), compared to a control dose quantified and standardized to 2 mg/day of PACs on mean number of new UTIs during a 6-month follow-up period.

DETAILED DESCRIPTION:
Cranberry juice, fruit (fresh and dried), functional foods, and cranberry dietary supplements are promoted for prevention of urinary tract infections (UTIs) on the basis of their content of cranberry proanthocyanidins (PACs) with "A-type" interflavan bonds. Several clinical trials have assessed efficacy of cranberry-derived products, essentially with cranberry juices, but discordant results have been found. Lack of compliance but mostly lack of standardization in product concentrations can account for the variability among results. Indeed, most clinical trials do not report quantity of PACs. According to most recent studies, quantification of PACs requiring standardized and reproducible methods should be at least 37 mg/day. It can be hypothesized that efficacy of cranberry extract in UTIs prevention among young women can be strongly increased using optimal dosage (standardized to 37 mg/day of PACs). The purpose of this clinical trial study is to assess, among young and sexually active women presenting recurrent UTIs, efficacy of an optimal dose of cranberry extract quantified and standardized to 37 mg/day of PACs, compared to a control dose quantified and standardized to 2 mg/day of PACs on mean number of new UTIs during a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and sexually active women
* Aged between 18 to 45 years old
* Recurrence of 2 UTIs in the past 6 months or 3 in the past year
* Do not have consumed cranberry juice, polyphenols or antioxidant supplements in the last 2 weeks
* Internet access

Exclusion Criteria:

* Women who have personal history of acute or chronic renal failure
* Women who have personal history of urogenital system anomalies, urogenital tractus surgery or intestinal diseases causing malabsorption (e.g., Crohn and celiac diseases)
* Women who have personal history of kidney stones, taking anticoagulant medication or have taken anticoagulant medication in the last month
* Women presenting cranberry allergy or intolerance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mean number of urinary tract infections | Within a 6-month period

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, M.Sc., MD., Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Babar A, Moore L, Leblanc V, Dudonne S, Desjardins Y, Lemieux S, Bochard V, Guyonnet D, Dodin S. High dose versus low dose standardized cranberry proanthocyanidin extract for the prevention of recurrent urinary tract infection in healthy women: a double-blind randomized controlled trial. BMC Urol. 2021 Mar 23;21(1):44. doi: 10.1186/s12894-021-00811-w. PMID 33757474
- [Derived] Asma B, Vicky L, Stephanie D, Yves D, Amy H, Sylvie D. Standardised high dose versus low dose cranberry Proanthocyanidin extracts for the prevention of recurrent urinary tract infection in healthy women [PACCANN]: a double blind randomised controlled trial protocol. BMC Urol. 2018 May 2;18(1):29. doi: 10.1186/s12894-018-0342-7. PMID 29716563